CLINICAL TRIAL: NCT05545579
Title: Comparative Effects of Circuit Training and Trunk Stabilization Techniques on Speed, Power and Dynamic Balance in Basketball Players
Brief Title: Comparative Effects of Circuit Training and Trunk Stabilization Technique in Basketball Players
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/RCR&AHS/22/0405
Record Dates: First submitted 2022-09-15; First posted 2022-09-19 (Actual); Last update posted 2023-04-03 (Actual); Status verified 2023-03

CONDITIONS: Basketball Players

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- circuit training (Experimental): Circuit training consisted of 6 exercises, divided in 2 blocks (1st block contains ½ squats, bench press and pushups and 2nd block contains burpees, squat thrust and lunges) of 3 minutes.
  Interventions: Other: circuit trainng
- Trunk stabilization techniques (Experimental): The stabilization exercise group will repeat 6 exercises (Balance Ball with Pocket Knife, Reverse Crunch, Russian Return, Shuttle, Leg Lift, and Back extension) for 6 weeks. Lane agility drill, Sprint test, Vertical jump test, Star excursion test will used to evaluate outcomes
  Interventions: Other: trunk stabilization techniques

INTERVENTIONS:
Other: circuit trainng — Circuit training consisted of 6 exercises, divided in 2 blocks (1st block contains ½ squats, bench press and pushups and 2nd block contains burpees, squat thrust and lunges) of 3 minutes. The stabilization exercise group will repeat 6 exercises (Balance Ball with Pocket Knife, Reverse Crunch, Russian Return, Shuttle, Leg Lift, and Back extension) for 6 weeks. Lane agility drill, Sprint test, Vertical jump test, Star excursion test will used to evaluate outcomes
  Arms: circuit training
Other: trunk stabilization techniques — The stabilization exercise group will repeat 6 exercises (Balance Ball with Pocket Knife, Reverse Crunch, Russian Return, Shuttle, Leg Lift, and Back extension) for 6 weeks. Lane agility drill, Sprint test, Vertical jump test, Star excursion test will used to evaluate outcomes
  Arms: Trunk stabilization techniques

SUMMARY:
In the sports world, physical training is the most important factor because physical training increases the efficiency and the effectiveness of the sports. The players performance depends on various factors, but the main factor of players performance is physical training. Training contributes tremendously towards the achievement of such aims of this area in sports. The circuit training is a non-stop, high intensity, basketball specific workout. It increases overall speed and quickness, explosive power, upper and lower body strength, vertical jump and, most of all, the athlete's conditioning.

DETAILED DESCRIPTION:
This study will be a randomized control trial and will be conducted in National stadium and Ravians Basketball club Lahore. The study will be completed within the time duration of six months. Non-probability convenience sampling technique will be used to collect the data. The sample size of total 24 athletes will be taken in this study. The participants will be divided into two groups i-e, one group will receive circuit training and other group will receive trunk stabilization exercises.

Circuit training consisted of 6 exercises, divided in 2 blocks (1st block contains ½ squats, bench press and pushups and 2nd block contains burpees, squat thrust and lunges) of 3 minutes. The stabilization exercise group will repeat 6 exercises (Balance Ball with Pocket Knife, Reverse Crunch, Russian Return, Shuttle, Leg Lift, and Back extension) for 6 weeks. Lane agility drill, Sprint test, Vertical jump test, Star excursion test will used to evaluate outcomes

ELIGIBILITY:
Inclusion Criteria:

* Males
* Age between 16-30 years
* No pain complaint
* Recreational activity
* Participate voluntarily
* Players have spent at least one year in sports

Exclusion Criteria:

* Higher BMI
* joint, meniscus, or ligament damage
* lower extremity surgical history
* persistent knee instability
* cardiac/musculoskeletal/vestibular/neurological issues

Ages: 16 Years to 30 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 24 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2023-10-15 (Estimated); Study Completion 2023-10-22 (Estimated)

PRIMARY OUTCOMES:
Agility test | 4 week
  The Agility T-Test is a popular test for determining how quickly athletes can go forward, backward, and side to side. The client must run 10 meters to point one, sidestep to point two, sidestep to point three, sidestep back to point one, then sprint back to the finish to complete the Agility T-Test. The procedure is then repeated, but in the other direction. From start to finish, each effort is timed and compared to established norms
Vertical jump test | 4 week
  The Vertical Jump test is used to evaluate a candidate's lower-body strength. A vertical jump test gauge is used to conduct the test. Applicants should stand with their feet level and hip width apart beneath the testing gauge, with their dominant side closer to the gauge. The person then raises their dominant arm and fingers vertically over their head.
  On the test gauge, the test assessor then set the applicant's reach height to zero (0). The leap must be done with both feet flat on the ground without taking a step or running up from the starting position. To safeguard their lower limbs, candidates must take off and land with both feet. Only two (2) tries are permitted for applicants who must leap 30cm or greater
Star excursion balance test | 4 week
  The SEBT (Standing Excursion Balance Test) evaluates postural control and dynamic balance. It is currently widely used as a clinical evaluation tool. SEBT necessitates a combination of lower extremity strength, flexibility, and balance. This test is useful in determining whether or not a lower extremity athlete is at danger of injury, as well as musculoskeletal disorders in the lower limb, following a training programmed that improves postural control

CONTACTS AND LOCATIONS:
Overall Officials: Amna Shahid, t-DPT, Principal Investigator — Riphah International University
Locations (1):
- Pakistan sports board, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No